CLINICAL TRIAL: NCT05725408
Title: Comparison of a Telehealth Versus In-person Intervention for Binge Eating Among Adults and Adolescents
Brief Title: Comparison of a Telehealth Versus In-person Intervention for Binge Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Psi Chi (Other); American Psychological Foundation (Other); Academy for Eating Disorders (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2022-0163D
Record Dates: First submitted 2023-01-18; First posted 2023-02-13 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-01

CONDITIONS: Binge Eating
Keywords: binge eating; body image disturbance; telehealth; feasibility
MeSH Terms: conditions — Bulimia | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either an in-person group or a telehealth group. Both will receive the same intervention but using different formats for delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Group (Experimental): Participants will be randomized to the telehealth group where they will attend weekly group intervention sessions online through the Zoom platform. Participants will be emailed or mailed materials for session since they will not be attending in-person. Participants will not be asked to attend any sessions or portions of the study in-person.
  Interventions: Behavioral: Dialectical behavior therapy-informed group eating intervention protocol (telehealth)
- In-Person Group (Active Comparator): Participants will be randomized to the in-person group where they will attend weekly group intervention sessions at a building on the Texas A&M University campus. Participants will be emailed or provided session materials when they arrive for sessions. After the first session, they will not be attending any online sessions.
  Interventions: Behavioral: Dialectical behavior therapy-informed group eating intervention protocol (in-person)

INTERVENTIONS:
Behavioral: Dialectical behavior therapy-informed group eating intervention protocol (telehealth) — A 10-week, skills-based group eating intervention. Online/telehealth meetings will last approximately 1 hour each session, besides the first session (1.5 hours, orientation and assessments) and the final session (approx. 2-2.5 hours, session plus final assessments and exit interview).
  Arms: Telehealth Group
Behavioral: Dialectical behavior therapy-informed group eating intervention protocol (in-person) — A 10-week, skills-based group eating intervention. In-person meetings will last approximately 1 hour each session, besides the first session (1.5 hours, orientation and assessments, online) and the final session (approx. 2-2.5 hours, session plus final assessments and exit interview).
  Arms: In-Person Group

SUMMARY:
Adults and adolescents will be asked to participate in a 10-week intervention to better understand their emotions and improve their relationship with food.

DETAILED DESCRIPTION:
Adults and adolescents will be asked to participate in a 10-week eating intervention to better understand and manage their emotions and improve their relationship with food. Participants will fill out questionnaires related to their engagement in body avoidance behaviors and disordered eating, and assess their self-reported levels of impulsivity, food insecurity, mindfulness skills, emotion regulation skills, and distress tolerance skills. Participants will also be asked questions to assess the feasibility and acceptability of the telehealth format.

ELIGIBILITY:
Inclusion Criteria for Adolescent Group:

* Adolescent in high school (ages ~13-18)
* Participant and their caregiver must be able to understand and speak English
* Has access to a computer device or tablet with a microphone and web camera
* Has access to a reliable internet connection and a private, quiet place to complete sessions
* Willing or able to secure transportation to the Texas A&M University campus if selected for the in-person group
* Engages in loss-of-control eating AND eating within a 2-hour period what most people would consider an unusually large amount of food given the circumstances

Exclusion Criteria for Adolescent Group:

* Active suicidal ideation within the past 2 weeks
* Has been diagnosed with an intellectual disability
* Active psychosis or experiencing psychosis symptoms
* Caregiver is not able to participate

Inclusion for Adult Group:

* Age 18+
* Speaks and understands English
* Has access to a computer device or tablet with a microphone and web camera
* Has access to a reliable internet connection and a private, quiet place to complete sessions
* Willing or able to secure transportation to the Texas A&M University campus if selected for the in-person group
* Engages in loss-of-control eating AND eating within a 2-hour period what most people would consider an unusually large amount of food given the circumstances

Exclusion Criteria for Adult Group:

* Active suicidal ideation within the past 2 weeks
* Has been diagnosed with an intellectual disability
* Active psychosis or experiencing psychosis symptoms

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Change in binge eating | Participants will be asked to complete a measure of binge eating at baseline and immediately after the last session of the intervention (Week 10) to assess change in binge eating behaviors.
  Episodes and frequency of binge eating and binge eating behaviors via the Eating Disorder Examination Questionnaire. Two items from this scale will be used to assess for the number of episodes and frequency of binge eating. Participants are asked to respond with numeric values to these items according to their subjective view (e.g., may write "8" to to represent eight episodes of binge eating over the past 28 days). Partcipants provide a numeric response from 0+ (no maximum number). Higher scores indicate more episodes of binge eating.
Feasibility of attending and engaging in a binge eating intervention. | Participants will be asked these questions via a brief exit interview immediately after the last session of the intervention (Week 10) to assess intervention feasibility.
  Participants will be asked open-ended questions in an interview format about the feasibility of attending and engaging in a binge eating intervention (telehealth or in-person). For example, one of the items asks, "Were there too many sessions or just enough?"
Satisfaction with the binge eating intervention | Participants will be asked questions immediately after the last session of the intervention (Week 10).
  Participants will be asked nine questions developed by the author and collaborators about how acceptable they found the intervention (telehealth or in-person) to be (e.g., "I would recommend this program to a friend or family member who has difficulty with binge eating"). Six of the questions can be answered with either "Yes", "No", or "Don't know." The remaining three items are open-ended.

SECONDARY OUTCOMES:
Change in body image avoidance | Participants will be asked to complete the Body Image Avoidance Questionnaire weekly to assess changes in body image avoidance throughout the intervention (at baseline/pre-intervention and every week at the beginning of the session, weeks 2-10).
  Engagement in body image avoidance behaviors (e.g., actively refraining from looking in the mirror) assessed via the Body Image Avoidance Questionnaire. Participants can respond according to a Likert scale of 1 (Rarely or Never) through 5 (Always). The total score can range from 0 to 95. Higher scores indicate greater body image avoidance.
Change in appearance overvaluation | Participants will be asked to complete the Beliefs About Appearance Scale weekly to assess change in appearance overvaluation throughout the intervention (at baseline and every week at the beginning of the session, weeks 2-10).
  The extent to which participants place large value on their appearance assessed via the Beliefs About Appearance Scale. Participants can respond according to a Likert scale of 0 (Not at all) to 4 (Extremely). Higher scores indicate greater appearance overvaluation.
Change in disordered eating (other than binge eating) | Participants will be asked to complete a measure of disordered eating at baseline/pre-intervention and immediately after the final session of the intervention (Week 10).
  Engagement in behaviors representative of disordered eating (e.g., restriction of diet, excessive exercise, etc.) assessed via the Eating Disorder Examination Questionnaire. Most of the questions are answered by responding to a 7-point Likert scale ranging from 0 (No days) to 6 (Every day). Other items require a response in a numeric value provided by the participant (e.g., "6" for "6 days"). Other items require a response using a 7-point Likert scale ranging from 1 (Not at all) to 6 (Markedly). Participants who identify as "female" are also asked an additional question where they can either mark "yes" or "no." In all cases, positive or higher scores indicate greater engagement in disordered eating.
Change in impulsivity | Participants will be asked to complete a measure of impulsivity at baseline/pre-intervention and immediately after the final session of the intervention (Week 10).
  Engagement in impulsive behaviors (e.g., sensation-seeking) assessed via the UPPS-P Impulsive Behavior Scale (UPPS-P = urgency, premeditation, perseverance, sensation seeking, and positive urgency...it is not usually spelled out). Participants are asked to respond using a 4-point Likert scale ranging from 0 (Agree strongly) to 3 (Disagree strongly). Higher scores indicate higher levels of impulsivity.
Change in mindfulness skills | Participants will be asked to complete a measure of mindfulness at baseline/pre-intervention and immediately after the final session of the intervention (Week 10).
  Current engagement in mindful activities or practices assessed via the Kentucky Inventory of Mindfulness Skills. Participants are asked to respond using a 5-point Likert scale ranging from 1 (Never or very rarely true) to 5 (Very often or always true). Higher scores indicate more, or greater, use of mindfulness skills.
Change in emotion regulation | Participants will be asked to complete a measure of emotion regulation at baseline/pre-intervention and immediately after the final session of the intervention (Week 10).
  Ability to regulate or suppress emotions or engage in cognitive reappraisal are assessed via the Emotion Regulation Questionnaire (ERQ). Participants are asked to respond according to a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate greater use of cognitive reappraisal and emotional suppression.
Change in distress tolerance | Participants will be asked to complete a measure of distress tolerance at baseline and post-intervention (during the final group session).
  Ability to tolerate distress assessed via the Distress Tolerance Scale (DTS). Participants are asked to respond according to a 5-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). Higher scores indicate greater, or higher, distress tolerance.
Food insecurity | Participants will be asked to complete a measure of food insecurity at baseline/pre-intervention.
  Level of food insecurity assessed via the United States Household Food Security Survey Module: Six-item Short Form. Items are multiple choice (e.g., "often true", "sometimes true", "never true", or "don't know or refuse to answer"). Scores are coded and then scored such that higher scores indicate greater, or higher, food insecurity. Scores can range from 0 to 6.
Change in binge eating disorder status | Participants will be asked to complete a diagnostic measure of binge eating disorder at baseline/pre-intervention and immediately after the final session of the intervention (Week 10).
  The Questionnaire on Weight and Eating Patterns, Revised, Diagnostic and Statistical Manual of Mental Disorders Version 5 (QEWP-5) will be used to assess and diagnose individuals with binge eating disorder. Items are assessed using multiple choice and open-ended questions. Scores are summed together to determine whether the criteria for binge eating disorder are met.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT05725408/ICF_000.pdf